CLINICAL TRIAL: NCT03257423
Title: Acute Appendicitis and Microbiota - Ethology of Appendicitis and Effects of the Antimicrobial Treatment - The MAPPAC (Microbiology Appendicitis Acuta) Trial
Brief Title: Acute Appendicitis and Microbiota - Etiology of Appendicitis and Antibiotic Therapy Effects
Acronym: MAPPAC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Turku University Hospital (Other Government)
Collaborators: Tampere University Hospital (Other); Oulu University Hospital (Other); Kuopio University Hospital (Other); Helsinki University Central Hospital (Other); Jyväskylä Central Hospital (Other)
Responsible Party: Principal Investigator, Paulina Salminen, MD, PhD, Chief of Acute Care Surgery, Turku University Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: MAPPAC
Record Dates: First submitted 2017-08-02; First posted 2017-08-22 (Actual); Last update posted 2020-11-10 (Actual); Status verified 2020-11

CONDITIONS: Acute Appendicitis
Keywords: Uncomplicated acute appendicitis; Complicated acute appendicitis; Antibiotic therapy; Microbiological etiology
MeSH Terms: conditions — Appendicitis | interventions — Metronidazole; Moxifloxacin; Appendectomy

STUDY DESIGN:
Intervention Model Description: Patients are enrolled in conjuction with APPAC II (NCT03236961) and APPAC III (NCT 03234296) trials, all patients with uncomplicated or complicated acute appendicitis are evaluated for MAPPAC enrollment. MAPPAC study groups: complicated acute appendicitis (samples: rectal swabs, serum, removed appendix), APPAC II patients in two groups according to APPAC II randomized antibiotic therapy (uncomplicated acute appendicitis, samples: rectal swabs, serum and in cases of antibiotic treatment failure or appendicitis recurrence also removed appendix), APPAC III patients in two groups according to APPAC III randomized group of antibiotc or placebo therapy (uncomplicated acute appendicitis, samples: rectal swabs, serum and in cases of antibiotic or placebo treatment failure or appendicitis recurrence also removed appendix), and patients with uncomplicated acute appendicitis declining to participate in APPAC II or III trials undergoing appendectomy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- I.v. + p.o. antibiotics (APPAC II) (Active Comparator): Patients in this group recruited also in APPAC II trial will receive i.v. antibiotics (ertapenem 1 g twice per day) for 2 days followed by p.o. antibiotics (levofloxacin 500 mg x 1 and metronidazole 500 mg x 3) for 5 days, for a total treatment duration of 7 days. From these patients, rectal swab samples will be collected at day 0 (before treatment) and day 1 (after beginning of treatment), serum sample before treatment initiation.
  Interventions: Drug: Ertapenem followed by levofloxacin and metronidazole
- P.o. moxifloxacin (APPAC II) (Active Comparator): Patients in this group recruited also in APPAC II trial will receive p.o. antibiotics for a total of 7 days, moxifloxacin 400 mg once per day. From these patients, rectal swab samples of faces will be collected at two time points, day 0 (before treatment) and day 1 (after beginning of treatment), serum sample before treatment initiation.
  Interventions: Drug: Moxifloxacin
- Placebo treatment (APPAC III) (Placebo Comparator): Patients in this group recruited also in APPAC III trial will receive i.v. placebo 3 times per day for 3 days followed by p.o. placebo 3 times per day for 4 additional days. From these patients rectal swab samples will be collected twice during the stay at the research hospital (time points 0 and 1 or 3 d) and three times at home (follow-up at one week, six months and one year). Serum samples are taken prior to treatment initiation and at 10 days after the treatment initiation.
  Interventions: Other: Placebo
- Surgery (complicated appendicitis) (Other): Patients in this group will undergo appendectomy and are recruited only in the MAPPAC trial. Rectal swab samples and biopsies from the removed appendix will be collected from these patients.
  Interventions: Procedure: Appendectomy
- Surgery (uncomplicated appendicitis) (Other): Patients in this group will undergo appendectomy either after refusing to participate in the APPAC II or APPAC III trials or after presenting with recurrent appendicitis after antibiotic or placebo therapy. Rectal swab samples of faces and biopsies from the removed appendix will be collected from these patients.
  Interventions: Procedure: Appendectomy
- I.v. + p.o. antibiotics (APPAC III) (Active Comparator): Patients in this group recruited also in APPAC III trial will receive i.v. antibiotics (ertapenem 1 g twice per day) for 3 days followed by p.o. antibiotics (levofloxacin 500 mg x 1 and metronidazole 500 mg x 3) for 4 days, for a total treatment duration of 7 days. From these patients rectal swab samples will be collected twice during the stay at the research hospital (time points 0 and 1 or 3 d) and three times at home (follow-up at one week, six months and one year). Serum samples are taken prior to treatment initiation and at 10 days after the treatment initiation.
  Interventions: Drug: Ertapenem followed by levofloxacin and metronidazole

INTERVENTIONS:
Drug: Ertapenem followed by levofloxacin and metronidazole — Ertapenem 1 g i.v. daily for either 2 days (MAPPAC + APPAC II patients) or 3 days (MAPPAC + APPAC III) followed by p.o. levofloxacin 500 mg x 1 + metronidazole 500 mg x 3 for either 5 days (APPAC II + MAPPAC) or 4 days (APPAC III + MAPPAC)
  Arms: I.v. + p.o. antibiotics (APPAC II); I.v. + p.o. antibiotics (APPAC III)
Drug: Moxifloxacin — Moxifloxacin 400 mg once a day for seven days (APPAC II + MAPPAC)
  Arms: P.o. moxifloxacin (APPAC II)
Procedure: Appendectomy — Primarily laparoscopic appendectomy for either complicated acute appendicitis or uncomplicated acute appendicitis (refusing to participate in APPAC II or III trials or recurrent acute appendicitis).
  Arms: Surgery (complicated appendicitis); Surgery (uncomplicated appendicitis)
Other: Placebo — Placebo i.v. once a day for three days (APPAC III + MAPPAC) followed by placebo capsules three times a day for four days.
  Arms: Placebo treatment (APPAC III)

SUMMARY:
Appendicectomy has been the treatment of acute appendicitis for over a hundred years. Appendicectomy, however, includes operative and postoperative risks despite being a routine procedure. Several studies have proved promising results of the safety and efficiency of antibiotics in the treatment of acute uncomplicated appendicitis. The previous APPAC study by the investigators, published in 2015 in the Journal of American Medical Association, also proved promising results with 73% of patients with uncomplicated appendicitis treated successfully with antibiotics. None of the patients initially treated with antibiotics that later had appendectomy had major complications. The results of the APPAC trial suggest that CT proven uncomplicated acute appendicitis is not a surgical emergency and antibiotic therapy is a safe first-line treatment option. Reducing unnecessary appendectomies has also been shown to lead to significant economic savings. On the other hand, antibiotic therapies have been shown to have an effect on the normal gut microbiota and are considered an increasing global health threat underlining the importance of evaluating both short- and long-term effects of the antimicrobial treatment in old and new indications.

The aims of this randomized prospective study are:

1. To evaluate the possible role and differences in the microbiological etiology of complicated and uncomplicated appendicitis.
2. To determine the effects of both antibiotic and placebo treatment on the composition of gut microbiota, and to evaluate how it recovers after the appendicitis-related antimicrobial treatment (AMT)
3. To evaluate the effects of the duration of the hospital stay on the AMR reservoir of the gut microbiota.

DETAILED DESCRIPTION:
Appendectomy has been the treatment of acute appendicitis for over a hundred years. Appendicectomy, however, includes operative and postoperative risks despite being a routine procedure. Several studies have proved promising results of the safety and efficiency of antibiotics in the treatment of acute uncomplicated appendicitis. The previous APPAC study by the investigators, published in 2015 in the Journal of American Medical Association, also proved promising results with 73% of patients with uncomplicated appendicitis treated successfully with antibiotics. None of the patients initially treated with antibiotics that later had appendectomy had major complications. The results of the APPAC trial suggest that CT proven uncomplicated acute appendicitis is not a surgical emergency and antibiotic therapy is a safe first-line treatment option. Reducing unnecessary appendectomies has also been shown to lead to significant economic savings. On the other hand, antibiotic therapies have been shown to have an effect on the normal gut microbiota.

Gut microbiota is an extremely complex ecosystem with both high bacterial density and diversity. Recent scientific evidence emphasizes that the symbiosis between the host and the balanced gut microbiota supports good health, and contributes to various biochemical and metabolic functions occurring in host's body. The possible role of the somehow distorted gut microbiota composition in addition to its metabolites in the etiopathogenesis of many diseases such as allergy, inflammatory bowel disease, type 1 diabetes and obesity related disorders, has been recently proposed. Further, detected alterations and perturbations both in the gut microbiota composition and functionality have been linked to the development of various malignancies such as colorectal cancer, gastric cancer and hepatocellular carcinoma. To date, the role of the microbes and especially the members of the commensal microbiota with their structural compartments and metabolites in the pathogenesis and etiology of appendicitis have not been clarified in detail, despite the recent knowledge that uncomplicated acute appendicitis could be treated by antibiotic treatments alone. Further, there is only limited amount of evidence on the appendix microbial composition in humans.

Microbial overgrowth has been speculated to serve as a secondary consequence in appendicitis. However, recent accumulating evidence suggests that primary bacterial infection may actually be an initiating event in the pathogenesis of the disease. Interestingly, it has been postulated that the appendix could serve as a microbial reservoir for repopulating the gastrointestinal tract in times of necessity thus gut microbiota may act as a source for these pathogenic intruders. Further it has been reported that certain members of the gram negative Fusobacteria especially F. nucleatum and necrophorum are present in most appendicitis samples.

Additionally, antimicrobial resistance (AMR) is considered an increasing global threat. According to the WHO (World Health Organisation), in 2050s more people will be killed by AMR bacteria than by all cancers.The use of antimicrobials in humans and especially in animal health care and production industry are the major causes of increasing AMR worldwide; the prudent use of antimicrobials is essential to prevent increasing AMR. Antimicrobials are known to decrease the gut microbiota diversity, richness and species variation and cause the perturbation of its overall balance and even a short-term antimicrobial treatment has a long-term impact on its composition underlining the importance of evaluating both short- and long-term effects of the antimicrobial treatment in old and new indications.

The aims of this randomized prospective study are:

1. To evaluate the possible role and differences in the microbiological etiology of complicated and uncomplicated appendicitis. The bacterial composition of the complicated appendix will be compared to the gut microbiota composition determined from the fecal sample collected from the same individual. Additionally, these results will be compared to the gut microbiota composition of patients with uncomplicated acute appendicitis.
2. To determine the effects of both antibiotic and placebo treatment on the composition of gut microbiota, and to evaluate how it recovers after the appendicitis-related antimicrobial treatment (AMT). The bacterial composition and AMR reservoir of the gut microbiota will be evaluated both pre and post treatment in patients receiving antibiotic or placebo treatment for uncomplicated acute appendicitis. Additionally, the recovery of gut microbiota composition and disappearance of AMR will be evaluated. We will compare two variations (i.v.and p.o.) of antibiotic treatment with the placebo treatment.
3. To evaluate the effects of the duration of the hospital stay on the AMR reservoir of the gut microbiota. According to the study protocols of the APPAC II and III trials, patients will spend either 1 or 3 days in the hospital in order to receive treatment before continuing the selected treatment at home. We will evaluate the effects of length of stay on the AMR reservoir of gut microbiota as well as evaluating if and when possible colonization occurs.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-60 years
* CT confirmed uncomplicated or complicated acute appendicitis
* Ability to give consent to participate in the study

Exclusion Criteria:

* Age under 18 years or over 60 years
* Pregnancy or lactation
* Allergy to contrast media or iodine
* Allergy or contraindication to antibiotic therapy
* Renal insufficiency
* Metformin medication
* Severe systemic illness (for example malignancy, medical condition requiring immunosuppressant medication)
* Inability to co-operate and give informed consent

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2017-04-04 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Microbiology in the etiology of acute appendicitis | 1 day
  Differences in the microbiological etiology of complicated and uncomplicated appendicitis

SECONDARY OUTCOMES:
Effects of antimicrobial treatment on gut microbiota | 1 year
  Determining the effects of both antibiotic and placebo treatment on the composition of gut microbiota, and to evaluate how it recovers after the appendicitis-related antimicrobial treatment evaluated by rectal swabs pre- and post treatment
Effects of hospital stay duration on the AMR reservoir of the gut microbiota | 3 days
  The effect of length of hospital stay (days) on the AMR reservoir of gut microbiota and colonization occurrence evaluated by analysing rectal swabs microbiota pre- and post-treatment at 0, 1 and 3 days.

CONTACTS AND LOCATIONS:
Overall Officials: Paulina Salminen, MD, PhD, Principal Investigator — Turku University Hospital
Locations (1):
- Turku University Hospital, Turku, Finland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Vanhatalo S, Makila E, Hakanen AJ, Munukka E, Salonen J, Saarinen T, Gronroos J, Sippola S, Salminen P. Appendicolith classification: physical and chemical properties of appendicoliths in patients with CT diagnosed acute appendicitis - a prospective cohort study. BMJ Open Gastroenterol. 2024 Aug 19;11(1):e001403. doi: 10.1136/bmjgast-2024-001403. PMID 39160081
- [Derived] Vanhatalo S, Munukka E, Kallonen T, Sippola S, Gronroos J, Haijanen J, Hakanen AJ, Salminen P. Appendiceal microbiome in uncomplicated and complicated acute appendicitis: A prospective cohort study. PLoS One. 2022 Oct 14;17(10):e0276007. doi: 10.1371/journal.pone.0276007. eCollection 2022. PMID 36240181
- [Derived] Vanhatalo S, Munukka E, Sippola S, Jalkanen S, Gronroos J, Marttila H, Eerola E, Hurme S, Hakanen AJ, Salminen P; APPAC collaborative study group. Prospective multicentre cohort trial on acute appendicitis and microbiota, aetiology and effects of antimicrobial treatment: study protocol for the MAPPAC (Microbiology APPendicitis ACuta) trial. BMJ Open. 2019 Sep 6;9(9):e031137. doi: 10.1136/bmjopen-2019-031137. PMID 31494621